CLINICAL TRIAL: NCT02873130
Title: Effectiveness of Telepractice by Smartphone App Technology in Preventing Voice Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Chester University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Elizabeth Grillo, Associate Professor, West Chester University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R15DC014566-01 (NIH)
Record Dates: First submitted 2016-08-08; First posted 2016-08-19 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Prevention of Voice Disorders in Student Teachers

ARMS (3):
- Behavioral: Telepractice Global Voice Prevention Model (Experimental): Participants will complete the Global Voice Prevention Model (GVPM) through West Chester University's Desire 2 Learn (D2L) software program. Synchronous and asynchronous learning opportunities are provided through D2L over a four week period. The GVPM includes vocal hygiene, vocal education, and vocal training.
  Interventions: Behavioral: Telepractice Global Voice Prevention Model
- Behavioral: In-person Global Voice Prevention Model (Experimental): Participants will complete the Global Voice Prevention Model (GVPM) at West Chester University in-person. The GVPM will meet for 2 hours once a week for four weeks. The GVPM includes vocal hygiene, vocal education, and vocal training.
  Interventions: Behavioral: In-person Global Voice Prevention Model
- Behavioral: Telepractice, Vocal Hygiene and Vocal Education (Sham Comparator): Participants will complete Vocal Hygiene and Vocal Education through West Chester University's Desire 2 Learn (D2L) software program. Asynchronous learning opportunities are provided through D2L over a one week period.
  Interventions: Behavioral: Telepractice, Vocal Hygiene and Vocal Education

INTERVENTIONS:
Behavioral: Telepractice Global Voice Prevention Model
  Arms: Behavioral: Telepractice Global Voice Prevention Model
Behavioral: In-person Global Voice Prevention Model
  Arms: Behavioral: In-person Global Voice Prevention Model
Behavioral: Telepractice, Vocal Hygiene and Vocal Education
  Arms: Behavioral: Telepractice, Vocal Hygiene and Vocal Education

SUMMARY:
Voice disorders in teachers have a significant impact on communication, quality of life, and economic costs to the healthcare system. We need to advance the prevention of voice disorders in teachers by testing an online telepractice model with synchronous (in real-time) and asynchronous (stored and accessed later) methods. The current study will investigate the effectiveness of the theoretically-driven Global Voice Prevention Model (GVPM) delivered by two methods; 1) online telepractice (synchronous and asynchronous) and 2) traditional, in-person for vocally healthy physical education and vocal music student teachers. Effectiveness of the model will be assessed by voice-related measures captured daily on a smartphone app during student teaching, matching the asynchronous aspects of the telepractice model and representing the effects of vocal loading from teaching.

ELIGIBILITY:
Inclusion Criteria:

* senior at West Chester University as of fall 2016 and fall 2017,
* student teaching during spring 2017 or 2018,
* healthy voice user,
* owns a smartphone

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Presence and frequency of a voice problem | AM (before teaching) and PM (after teaching) 5 days a week for up to 3 months.
  Question will be asked twice a day before and after teaching.

SECONDARY OUTCOMES:
Acoustic: fundamental frequency | AM (before teaching) and PM (after teaching) 5 days a week for up to 3 months.
  Participants will record sustained aaaahhh, we were away a year ago, and describe their voice for 15 seconds twice a day before and after teaching.
Acoustic: standard deviation of fundamental frequency | AM (before teaching) and PM (after teaching) 5 days a week for up to 3 months.
  Participants will record sustained aaaahhh, we were away a year ago, and describe their voice for 15 seconds twice a day before and after teaching.
Acoustic: jitter% | AM (before teaching) and PM (after teaching) 5 days a week for up to 3 months.
  Participants will record sustained aaaahhh, we were away a year ago, and describe their voice for 15 seconds twice a day before and after teaching.
Acoustic: shimmer% | AM (before teaching) and PM (after teaching) 5 days a week for up to 3 months.
  Participants will record sustained aaaahhh, we were away a year ago, and describe their voice for 15 seconds twice a day before and after teaching.
Acoustic: cepstral peak prominence | AM (before teaching) and PM (after teaching) 5 days a week for up to 3 months.
  Participants will record sustained aaaahhh, we were away a year ago, and describe their voice for 15 seconds twice a day before and after teaching.
Perceptual: Voice Handicap Index | AM (before teaching) and PM (after teaching) 5 days a week for up to 3 months.
  Quality of life questions.
Perceptual: Vocal Fatigue Index | AM (before teaching) and PM (after teaching) 5 days a week for up to 3 months.
  Vocal fatigue questions
Perceptual: perceptions of voice | AM (before teaching) and PM (after teaching) 5 days a week for up to 3 months.
  Perceptions of voice based on the Consensus-auditory Perceptual Evaluation of Voice.
Aerodynamic: sustained aaaaahhhhh | AM (before teaching) and PM (after teaching) 5 days a week for up to 3 months.
  Participants will say aaaaahhhh as long as they can to determine how well they are managing airflow with phonation twice a day before and after teaching.
Aerodynamic: s/z ratio | AM (before teaching) and PM (after teaching) 5 days a week for up to 3 months.
  Participants will say s and z as long as they can to determine how well they are managing airflow with phonation twice a day before and after teaching.

CONTACTS AND LOCATIONS:
Locations (1):
- Elizabeth Grillo, West Chester, Pennsylvania, United States